CLINICAL TRIAL: NCT01265940
Title: Target-specific Therapy With Pazopanib as Add-on to Vinflunine in Patients With Advanced or Metastatic Urothelial Carcinoma of the Bladder After Failure of Platinum-based Treatment
Brief Title: Pazopanib and Vinflunine in Urothelial Cancer of the Bladder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Thomas Otto (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Thomas Otto, Prof. Dr. Thomas Otto, Lukas-Krankenhaus GmbH
Organization: Lukas-Krankenhaus GmbH (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZITM1
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Advanced Urothelial Cancer of Bladder After Failure of Platinum-containing Therapy.
Keywords: bladder cancer; urothelial cancer; metastatic urothelial cancer; advanced urothelial cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pazopanib; vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib + Vinflunine (Experimental)
  Interventions: Drug: Pazopanib as add-on to vinflunine

INTERVENTIONS:
Drug: Pazopanib as add-on to vinflunine — Patients will receive vinflunine standard regimen (intravenous infusion every three weeks) as specified per drug label plus additional pazopanib as daily oral medication. Doses of pazopanib will be escalated in 200 mg/d steps during phase I up to a maximum of 800 mg/d.
  In Phase II the patients will be given pazopanib + vinflunine at maximum tolerated dose.
  Other Names: Pazopanib is marketed as Votrient.; Vinflunine is marketed as Javlor.

SUMMARY:
Urothelial carcinoma of the bladder mostly is chemically induced and represents the second prevalent urooncological disease. About 20% of newly diagnosed urothelial carcinoma cases of the bladder are already advanced or metastasized. Before 2008 2009 no second line therapy after failure of primary systemic therapy of advanced / metastatic disease was established outside of clinical trials. The actual standard for this situation was a supportive, symptomatic therapy. Vinflunine has demonstrated improved survival from 4.3 to 6.9 months (p=0.04), with an adequate disease control, good symptom control and with acceptable toxicity. Based on these results, this compound became standard se¬cond line treatment for refractory metastatic bladder cancer disease after failure of platinum-containing therapy. As the prognosis still remains poor, new treatment opportunities have to be explored.

The target-specific therapy with Pazopanib suggests a positive influence of both inductive and perioperative treatment of solid tumors. Pazopanib has been approved by the FDA and the EMA for the treatment of advance renal cell carcinoma. Results for advanced urothelial carcinoma are missing so far as well as data on tolerability of the combination of both vinflunine and pazopanib. As the pharmacodynamic properties as well as the safety profile of both drugs are different, assumption is justified that there might occur additive efficacy effects without addition of adverse outcomes. Aim of the study thus is

1. To define the maximum tolerated dose (MTD) of Pazopanib in combination with Vinflunine in a phase-I-setting and
2. To further assess efficacy and safety of the combination at the MTD level in phase II.

During the pase-I-part of the study different doses of pazopanib will be added to the standard vinflunine scheme in groups of 6 patients maximum. Dose escalation will only be performed in the next patient group if not more than one out of six patients shows dose-limiting toxicity. Each patient will be treated with the drug combination for a duration of two vinflunine cycles, that is six weeks.

During the phase-II study new patients will be treated with the drug combination at maximum-tolerated dose until disease progression (assessed by RECIST 1.1 procedures).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* Histologically confirmed Transitional Cell Carcinoma of the Urothelium (TCCU) with lymphatic (N-stage 2-3) and/or distant metastases (M-stage 1) not amenable to definitive regional/local therapy
* Progression of tumor disease after platinum containing systemic chemotherapy for advanced or metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 1
* estimated minimal life expectancy of 3 months at screening
* At least one measurable tumor lesion according to RECIST 1.1 criteria
* Adequate organ system function at screening
* Adequate contraception

Exclusion Criteria:

* More than 1 prior chemotherapy, biologic therapy or hormonal therapy within 14 days prior to the first dose of study medication
* Prior malignancy within 5 years prior to inclusion (exception: successfully treated basal cell carcinoma or in situ carcinoma)
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding within 28 days prior to beginning study treatment, e.g

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion/s with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product, e.g.

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel
* Active infection requiring antibiotics within 14 days before registration
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula at screening
* Screening-electrocardiogram (ECG) with any significant modifi¬cations suggesting a high risk of occurrence of an acute clinical event (such as signs of angina pectoris, high risk arrhythmia etc.)
* History of one or more of the following cardiac / cardiovascular conditions within the past 6 months before registration:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
  * NYHA Class II, III or IV congestive heart failure
  * Uncontrolled cardiac arrhythmia
* Poorly controlled hypertension, defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90 mmHg
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months before registration
* Peripheral neuropathy grade ≥ 2 (NCI CTC v3.0)
* Unstable diabetes mellitus
* Uncontrolled hypercalcaemia > 2.9 mmol/L
* Prior major surgery or trauma within 28 days prior to registration and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major)
* Evidence of active bleeding e.g. GI bleeding or bleeding diathesis at screening.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* Hemoptysis with bleeding of > 2.5 mL within 8 weeks before registration
* Any serious and/or unstable pre-existing medical, psychiatric/psychological, familial, sociological, geographical or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* prior to the first dose of study drug and for the duration of the study
* Radiation, surgery or tumor embolization or any investigational treatment within 14 days prior to the first dose of study medication
* Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or progressing in severity, except nausea, vomiting, alopecia
* ASA 4
* Pre-treatment with Pazopanib or Vinflunine
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Phase I: Definition of the Maximum Tolerated Dose (MTD) of Pazopanib in combination with Vinflunine. | 6 weeks (two cycles of vinflunine)
  MTD ist defined as the dose level with dose-limiting toxicity occurring in maximum one out of six patients.
Phase II: Progression-free survival rate | 3 months
  Progression-free survival will be assessed by means of RECIST 1.1. methodology

SECONDARY OUTCOMES:
Phase I: Progression-free survival rate, Phase II: Safety profile, overall survival | Six weeks after first administration of study drug.
  Progression-free survival will be assessed by means of RECIST 1.1. methodology

CONTACTS AND LOCATIONS:
Locations (1):
- Lukaskrankenhaus, Neuss, Germany